CLINICAL TRIAL: NCT00398931
Title: A 5-year, Double-blind, Randomized, Placebo-controlled Extension Study to Examine the Long-term Safety and Efficacy of Oral Alendronate in Postmenopausal Women Who Previously Received Alendronate in Conjunction With the Fracture Intervention Trial
Brief Title: FLEX - Long-term Extension of FIT (Fracture Intervention Trial)(0217-051)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-051; 2006_558
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217, alendronate sodium / Duration of Treatment : 5 Years
Drug: Comparator : placebo (unspecified) /Duration of Treatment : 5 Years

SUMMARY:
This study was conducted among women who had previously received alendronate for 3 to 6 years during the Fracture Intervention Trial (FIT). Participants in the FLEX study were randomly assigned to receive alendronate (either 5 or 10 mg/day) or matching placebo during the next 5 years, in order to evaluate the effects of continuing or discontinuing alendronate treatment on bone mineral density and biochemical markers of bone turnover.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, women needed to have previously participated in the Fracture Intervention Trial (FIT) and to have been part of the group treated with alendronate in FIT
* They needed to have received at least 3 years of treatment with alendronate in the FIT trial
* In addition, their bone mineral density (BMD) at the hip needed to be better than it was at the start of FIT

Exclusion Criteria:

* Patients were excluded if they had conditions that contraindicated alendronate therapy and if they might have used other medications for the treatment of osteoporosis
* Women were also excluded if BMD at the hip was below a certain level (T-score <=-3.5); that is, if it were 3.5 standard deviations or more lower than the average for young adult women

Ages: 60 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 1998-02; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Total hip bone mineral density (BMD)

SECONDARY OUTCOMES:
BMD of femoral neck, trochanter, and lumbar spine
Biochemical markers of bone turnover

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Black DM, Schwartz AV, Ensrud KE, Cauley JA, Levis S, Quandt SA, Satterfield S, Wallace RB, Bauer DC, Palermo L, Wehren LE, Lombardi A, Santora AC, Cummings SR; FLEX Research Group. Effects of continuing or stopping alendronate after 5 years of treatment: the Fracture Intervention Trial Long-term Extension (FLEX): a randomized trial. JAMA. 2006 Dec 27;296(24):2927-38. doi: 10.1001/jama.296.24.2927. PMID 17190893
- [Background] Black DM, Cummings SR, Karpf DB, Cauley JA, Thompson DE, Nevitt MC, Bauer DC, Genant HK, Haskell WL, Marcus R, Ott SM, Torner JC, Quandt SA, Reiss TF, Ensrud KE. Randomised trial of effect of alendronate on risk of fracture in women with existing vertebral fractures. Fracture Intervention Trial Research Group. Lancet. 1996 Dec 7;348(9041):1535-41. doi: 10.1016/s0140-6736(96)07088-2. PMID 8950879
- [Background] Bauer DC, Black D, Ensrud K, Thompson D, Hochberg M, Nevitt M, Musliner T, Freedholm D. Upper gastrointestinal tract safety profile of alendronate: the fracture intervention trial. Arch Intern Med. 2000 Feb 28;160(4):517-25. doi: 10.1001/archinte.160.4.517. PMID 10695692
- [Background] Black DM, Thompson DE, Bauer DC, Ensrud K, Musliner T, Hochberg MC, Nevitt MC, Suryawanshi S, Cummings SR; Fracture Intervention Trial. Fracture risk reduction with alendronate in women with osteoporosis: the Fracture Intervention Trial. FIT Research Group. J Clin Endocrinol Metab. 2000 Nov;85(11):4118-24. doi: 10.1210/jcem.85.11.6953. PMID 11095442
- [Background] Levis S, Quandt SA, Thompson D, Scott J, Schneider DL, Ross PD, Black D, Suryawanshi S, Hochberg M, Yates J; FIT Research Group. Alendronate reduces the risk of multiple symptomatic fractures: results from the fracture intervention trial. J Am Geriatr Soc. 2002 Mar;50(3):409-15. doi: 10.1046/j.1532-5415.2002.50102.x. PMID 11943033
- [Background] Bauer DC, Black DM, Garnero P, Hochberg M, Ott S, Orloff J, Thompson DE, Ewing SK, Delmas PD; Fracture Intervention Trial Study Group. Change in bone turnover and hip, non-spine, and vertebral fracture in alendronate-treated women: the fracture intervention trial. J Bone Miner Res. 2004 Aug;19(8):1250-8. doi: 10.1359/JBMR.040512. Epub 2004 May 24. PMID 15231011
- [Background] Cummings SR, Palermo L, Browner W, Marcus R, Wallace R, Pearson J, Blackwell T, Eckert S, Black D. Monitoring osteoporosis therapy with bone densitometry: misleading changes and regression to the mean. Fracture Intervention Trial Research Group. JAMA. 2000 Mar 8;283(10):1318-21. doi: 10.1001/jama.283.10.1318. PMID 10714731
- [Background] Cummings SR, Black DM, Thompson DE, Applegate WB, Barrett-Connor E, Musliner TA, Palermo L, Prineas R, Rubin SM, Scott JC, Vogt T, Wallace R, Yates AJ, LaCroix AZ. Effect of alendronate on risk of fracture in women with low bone density but without vertebral fractures: results from the Fracture Intervention Trial. JAMA. 1998 Dec 23-30;280(24):2077-82. doi: 10.1001/jama.280.24.2077. PMID 9875874
- [Background] Cauley JA, Thompson DE, Ensrud KC, Scott JC, Black D. Risk of mortality following clinical fractures. Osteoporos Int. 2000;11(7):556-61. doi: 10.1007/s001980070075. PMID 11069188
- [Background] Ensrud KE, Barrett-Connor EL, Schwartz A, Santora AC, Bauer DC, Suryawanshi S, Feldstein A, Haskell WL, Hochberg MC, Torner JC, Lombardi A, Black DM; Fracture Intervention Trial Long-Term Extension Research Group. Randomized trial of effect of alendronate continuation versus discontinuation in women with low BMD: results from the Fracture Intervention Trial long-term extension. J Bone Miner Res. 2004 Aug;19(8):1259-69. doi: 10.1359/JBMR.040326. Epub 2004 Mar 29. PMID 15231012
- [Background] Nevitt MC, Ross PD, Palermo L, Musliner T, Genant HK, Thompson DE. Association of prevalent vertebral fractures, bone density, and alendronate treatment with incident vertebral fractures: effect of number and spinal location of fractures. The Fracture Intervention Trial Research Group. Bone. 1999 Nov;25(5):613-9. doi: 10.1016/s8756-3282(99)00202-1. PMID 10574584
- [Background] Hochberg MC, Ross PD, Black D, Cummings SR, Genant HK, Nevitt MC, Barrett-Connor E, Musliner T, Thompson D. Larger increases in bone mineral density during alendronate therapy are associated with a lower risk of new vertebral fractures in women with postmenopausal osteoporosis. Fracture Intervention Trial Research Group. Arthritis Rheum. 1999 Jun;42(6):1246-54. doi: 10.1002/1529-0131(199906)42:63.0.CO;2-U. PMID 10366118
- [Background] Hochberg MC, Thompson DE, Black DM, Quandt SA, Cauley J, Geusens P, Ross PD, Baran D; FIT Research Group. Effect of alendronate on the age-specific incidence of symptomatic osteoporotic fractures. J Bone Miner Res. 2005 Jun;20(6):971-6. doi: 10.1359/JBMR.050104. Epub 2005 Jan 18. PMID 15883637
- [Background] Nevitt MC, Thompson DE, Black DM, Rubin SR, Ensrud K, Yates AJ, Cummings SR. Effect of alendronate on limited-activity days and bed-disability days caused by back pain in postmenopausal women with existing vertebral fractures. Fracture Intervention Trial Research Group. Arch Intern Med. 2000 Jan 10;160(1):77-85. doi: 10.1001/archinte.160.1.77. PMID 10632308
- [Background] Hochberg MC, Greenspan S, Wasnich RD, Miller P, Thompson DE, Ross PD. Changes in bone density and turnover explain the reductions in incidence of nonvertebral fractures that occur during treatment with antiresorptive agents. J Clin Endocrinol Metab. 2002 Apr;87(4):1586-92. doi: 10.1210/jcem.87.4.8415. PMID 11932287
- [Background] Ensrud KE, Thompson DE, Cauley JA, Nevitt MC, Kado DM, Hochberg MC, Santora AC 2nd, Black DM. Prevalent vertebral deformities predict mortality and hospitalization in older women with low bone mass. Fracture Intervention Trial Research Group. J Am Geriatr Soc. 2000 Mar;48(3):241-9. doi: 10.1111/j.1532-5415.2000.tb02641.x. PMID 10733048
- [Background] Papapoulos SE, Quandt SA, Liberman UA, Hochberg MC, Thompson DE. Meta-analysis of the efficacy of alendronate for the prevention of hip fractures in postmenopausal women. Osteoporos Int. 2005 May;16(5):468-74. doi: 10.1007/s00198-004-1725-z. Epub 2004 Sep 21. PMID 15448985
- [Background] Vogt TM, Ross PD, Palermo L, Musliner T, Genant HK, Black D, Thompson DE. Vertebral fracture prevalence among women screened for the Fracture Intervention Trial and a simple clinical tool to screen for undiagnosed vertebral fractures. Fracture Intervention Trial Research Group. Mayo Clin Proc. 2000 Sep;75(9):888-96. doi: 10.4065/75.9.888. PMID 10994823
- [Background] Quandt SA, Thompson DE, Schneider DL, Nevitt MC, Black DM; Fracture Intervention Trial Research Group. Effect of alendronate on vertebral fracture risk in women with bone mineral density T scores of-1.6 to -2.5 at the femoral neck: the Fracture Intervention Trial. Mayo Clin Proc. 2005 Mar;80(3):343-9. doi: 10.4065/80.3.343. PMID 15757015
- [Result] Schwartz AV, Bauer DC, Cummings SR, Cauley JA, Ensrud KE, Palermo L, Wallace RB, Hochberg MC, Feldstein AC, Lombardi A, Black DM; FLEX Research Group. Efficacy of continued alendronate for fractures in women with and without prevalent vertebral fracture: the FLEX trial. J Bone Miner Res. 2010 May;25(5):976-82. doi: 10.1002/jbmr.11. PMID 20200926
- [Result] Bauer DC, Schwartz A, Palermo L, Cauley J, Hochberg M, Santora A, Cummings SR, Black DM. Fracture prediction after discontinuation of 4 to 5 years of alendronate therapy: the FLEX study. JAMA Intern Med. 2014 Jul;174(7):1126-34. doi: 10.1001/jamainternmed.2014.1232. PMID 24798675